CLINICAL TRIAL: NCT03300180
Title: Caregiver Outcomes of Alzheimer's Disease Screening
Acronym: COADS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Nicole R. Fowler, PhD, Scientist, Indiana University Center for Aging Research, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 1705649205; 5R01AG056325-05 (NIH)
Record Dates: First submitted 2017-08-08; First posted 2017-10-03 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The patients in this group will receive no AD screening
- Screening Only (Active Comparator): The patients in this group will receive screening for AD. Patients and family members will receive a letter about how the patient performed on the screening. If they screen positive (e.g. ≤5 on the MIS-T or ≤2 on the Mini-Cog), the patient and family member will receive an infographic and some information about local clinical resources for them to peruse regarding follow-up care. The patient's PCP is also be notified of the screening results via EHR message.
  Interventions: Other: Screening Only
- Collaborative Dementia Care Program (Experimental): The patients in this group will receive screening for AD, Patients and family members will receive a letter about how the patient performed on the screening. If they screen positive (e.g. ≤5 on the MIS-T or ≤2 on the Mini-Cog), the patient and family member will receive an infographic. Also, the family member will receive two follow-up phone calls. One from the COADS Study Coordinator and one from a care coordinator at the Aging Brain Care Program (ABC). This phone call will include an opportunity for the family to ask questions and a conversation about the program and diagnostic evaluation and management. Dyads have the option to refuse the follow-up visit. The patient's PCP is also be notified of the screening results via EHR message,
  Interventions: Behavioral: Collaborative Dementia Care Program

INTERVENTIONS:
Behavioral: Collaborative Dementia Care Program — Much of the intervention, facilitated by care coordinator, is targeted to co-manage or support the practice behavior of primary care clinicians, enhance self-management skills of both the care-recipient and the informal caregiver, and maximize the coping behavior of the patient and the informal caregiver.
  Arms: Collaborative Dementia Care Program
Other: Screening Only — The patients in this group will receive screening for AD coupled with letters sent to the dyads and the primary care PCP informing them of the results of the screening
  Arms: Screening Only

SUMMARY:
This study will measure the risks and benefits of early screening of Alzheimer's disease. Early diagnosis through screening may enhance the family member's transition to a family caregiver and reduce caregiver burden by providing an opportunity for the family member to learn about the syndrome, receive interventions, and to prepare for their new care giving role.

DETAILED DESCRIPTION:
We are proposing the first randomized controlled trial (RCT) to evaluate the benefits and harms of AD screening on family members of older adults. The proposed trial will randomize 1,800 dyads (older adult and family member) into three groups. Older adults in the first group will be screened for AD at baseline coupled with disclosure of the screening results to the dyad and to the patient's primary care provider (Screening Only Group). Older adults in the second group will be screened for AD at baseline coupled with disclosure of the screening results and, if they screen positive, referred to the Aging Brain Care (ABC) Program for diagnostic evaluation and care, if AD is diagnosed (Screening Plus Group). Older adults in the third group will not be screened at baseline and will observed through surveillance of the patients' EHR for any screening or incident AD diagnoses that occurs as part of routine care. At the last follow-up assessment (24 months) we will we will screen the older adults and conduct an interview with the family caregiver to detect possible cognitive impairment (Control Group).

Specific Aim 1: Evaluate the impact of AD screening on family members' quality of life.

Hypothesis 1: In comparison to the control group, family members randomized to the screening only or the screening plus groups will express higher levels of health-related quality of life at 24 months as measured by the Short Form Health Survey (SF-36).

Specific Aim 2: Evaluate the impact of AD screening on family members' mood and anxiety.

Hypothesis 2: In comparison to the control group, family members randomized to the screening only or the screening plus groups will express lower rates of depressive and anxiety symptoms at 24 months as measured by the Patient Health Questionnaire (PHQ-9) and the Generalized Anxiety Disorder Scale (GAD-7).

Specific Aim 3: Assess the impact of AD screening on family members' caregiving preparedness and caregiving self-efficacy.

Hypothesis 3: In comparison to the control group, family members randomized to the screening only or the screening plus group, will be more prepared for caregiving and have higher self-efficacy at 24 months as measured by the Preparedness for Caregiving Scale and the Revised Scale for Caregiving Self-Efficacy.

Specific Aim 4: Compare the effectiveness of two strategies for diagnostic evaluation and management after AD screening.

Hypothesis 4: In comparison to the screening only group, family members randomized to the screening plus group will express higher levels of health-related quality of life, caregiver preparedness and caregiving self-efficacy and lower levels of depressive and anxiety symptoms at 24 months, as measured by the SF-36, Preparedness for Caregiving Scale, the Revised Scale for Caregiving Self-Efficacy, PHQ-9, and GAD-7, respectively.

ELIGIBILITY:
Inclusion Criteria:

Patients

* 65 years or older
* At least one visit to primary care practice within past 24 months
* Ability to provide informed consent
* Ability to communicate in English

Family Members

* 21 years or older
* Identified by the patient as the person most likely to provide them care if needed.*
* Lives with the patient or lives within a 50 mile radius.
* Ability to provide informed consent.
* Ability to communicate in English

Exclusion Criteria:

Patients

* Has a diagnosis of AD as determined by ICD-10 code.
* Evidence of a prescription for a cholinesterase inhibitors or memantine.
* Has serious mental illness such as bipolar or schizophrenia as determined by ICD-10 code
* Permanent resident of a nursing facility
* Already seen by the Healthy Aging Brain Care Program

Family Member

* Is a non-family member who is not a legal Healthcare Power of Attorney
* Has serious mental illness such as bipolar or schizophrenia as determined by ICD-10 code
* Has a diagnosis of AD as determined by ICD-10 code.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1822 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Fowler, PHD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Eskenazi Hospital, Indianapolis, Indiana
  - IU Health-Primary Care Clinics, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fowler NR, Head KJ, Perkins AJ, Gao S, Callahan CM, Bakas T, Suarez SD, Boustani MA. Examining the benefits and harms of Alzheimer's disease screening for family members of older adults: study protocol for a randomized controlled trial. Trials. 2020 Feb 19;21(1):202. doi: 10.1186/s13063-019-4029-5. PMID 32075686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dyads recruited in primary care clinic or over the phone.
Pre-assignment Details: Consented Dyads, consisting of patient and chosen family member. Randomization was completed after patient baseline to determine screening group arm.
Period: Baseline
Arm/Group | Control | Screening Only | Collaborative Dementia Care Program
Started | 608 (608 Patients and 608 Family members) | 607 (607 Patients and 607 Family member) | 607 (607 Patient and 607 Family member)
Completed (Due to intent to treat protocol a dyad will continue on in the study even if one or both miss an assessment. A death or withdrawal would remove both patient and family member of the dyad from continuing participation.) | 604 (604 Patients and 604 Family members- excluding those who withdrew after randomization) | 601 (601 Patients and 601 Family members- excluding those who withdrew after randomization) | 603 (603 Patients and 603 Family members excluding those who withdrew after randomization)
Not Completed | 4 | 6 | 4
Not completed — Withdrawal by Subject | 4 | 6 | 4
Period: 6 Month Outcome
Arm/Group | Control | Screening Only | Collaborative Dementia Care Program
Started (Each outcome will include previous completed participants and those missing due to intent to treat protocol.) | 604 (604 Patients and 604 Family members) | 601 (601 Patients and 601 Family members) | 603 (603 Patients and 603 Family members)
Completed (Due to intent to treat protocol a dyad will continue on in the study even if one or both miss an assessment. A death or withdrawal would remove both patient and family member of the dyad from continuing participation.) | 547 (547 Patients and 524 Family members) | 533 (533 Patients and 517 Family members) | 535 (535 Patients and 519 Family members)
Not Completed | 57 | 68 | 68
Not completed — Withdrawal by Subject | 12 | 12 | 19
Not completed — Death | 2 | 4 | 3
Not completed — Missed Assessment | 43 | 52 | 46
Period: 12 Month Outcome
Arm/Group | Control | Screening Only | Collaborative Dementia Care Program
Started (Each outcome will include previous completed participants and those missing due to intent to treat protocol.) | 590 (590 Patients and 590 Family members) | 585 (585 Patients and 585 Family members) | 581 (581 Patients and 581 Family members)
Completed (Due to intent to treat protocol a dyad will continue on in the study even if one or both miss an assessment. A death or withdrawal would remove both patient and family member of the dyad from continuing participation.) | 516 (516 Patients and 500 Family members) | 514 (514 Patients and 500 Family members) | 511 (511 Patients and 490 Family members)
Not Completed | 74 | 71 | 70
Not completed — Withdrawal by Subject | 3 | 6 | 6
Not completed — Death | 9 | 6 | 6
Not completed — Missed Assessment | 62 | 59 | 58
Period: 18 Month Outcome Assessment
Arm/Group | Control | Screening Only | Collaborative Dementia Care Program
Started (Each outcome will include previous completed participants and those missing due to intent to treat protocol.) | 578 (578 Patients and 578 Family members) | 573 (573 Patients and 573 Family members) | 571 (571 Patients and 571 Family members)
Completed (Due to intent to treat protocol a dyad will continue on in the study even if one or both miss an assessment. A death or withdrawal would remove both patient and family member of the dyad from continuing participation.) | 507 (507 Patients and 484 Family members) | 503 (503 Patients and 476 Family members) | 509 (509 Patients and 492 Family members)
Not Completed | 71 | 70 | 62
Not completed — Withdrawal by Subject | 14 | 4 | 13
Not completed — Death | 8 | 5 | 5
Not completed — Missed Assessment | 49 | 61 | 44
Period: 24 Month Outcome Assessment
Arm/Group | Control | Screening Only | Collaborative Dementia Care Program
Started (Each outcome will include previous completed participants and those missing due to intent to treat protocol.) | 556 (556 Patients and 556 Family members) | 564 (564 Patients and 564 Family members) | 553 (553 Patients and 553 Family members)
Completed (Due to intent to treat protocol a dyad will continue on in the study even if one or both miss an assessment. A death or withdrawal would remove both patient and family member of the dyad from continuing participation.) | 520 (520 Patients and 505 Family members) | 520 (520 Patients and 503 Family members) | 508 (508 Patients and 496 Family members)
Not Completed | 36 | 44 | 45
Not completed — Withdrawal by Subject | 6 | 10 | 4
Not completed — Death | 13 | 13 | 3
Not completed — Missed Assessment | 17 | 21 | 38

BASELINE CHARACTERISTICS:
Population: Baseline Demographic and Clinical Characteristics of Randomized Dyads, total unique participants aggregated by Patients and Family within each arm. Excluding Dyads who withdrew at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Screening Only | Collaborative Dementia Care Program | Total
Number analyzed (Participants) | 1208 | 1202 | 1206 | 3616
Age, Continuous [Mean (Standard Deviation); unit: years] — Patient characteristic: Patient Age Population: Patient Age,
  years
    number analyzed (Participants) | 604 | 601 | 603 | 1808
    (all) | 73.7 (5.7) | 73.5 (5.5) | 73.8 (5.8) | 73.7001 (5.701)
Age, Continuous [Mean (Standard Deviation); unit: in years] — Family Member Characteristic - Family Member Age Population: Family Member Age
  in years
    number analyzed (Participants) | 604 | 601 | 603 | 1808
    (all) | 63.8 (13.0) | 64.4 (12.7) | 64.4 (13.1) | 64.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Patient characteristic- Patient Sex Population: Patient Sex
  Participants
    number analyzed (Participants) | 604 | 601 | 603 | 1808
    Female | 338 | 318 | 303 | 959
    Male | 266 | 283 | 300 | 849
Sex: Female, Male [Count of Participants; unit: Participants] — Family Member Characteristic - Family Member Sex Population: Family Member Sex- excluding refused/withdrawn
  Participants
    number analyzed (Participants) | 604 | 601 | 602 | 1807
    Female | 406 | 407 | 411 | 1224
    Male | 198 | 194 | 191 | 583
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Patient characteristic- Patient Race/Ethnicity Population: Patient Race/Ethnicity
  Participants
    Asian: number analyzed (Participants) | 604 | 601 | 603 | 1808
    Asian | 4 | 8 | 3 | 15
    Black or African American: number analyzed (Participants) | 604 | 601 | 603 | 1808
    Black or African American | 92 | 81 | 67 | 240
    White: number analyzed (Participants) | 604 | 601 | 603 | 1808
    White | 505 | 506 | 525 | 1536
    Other: number analyzed (Participants) | 604 | 601 | 603 | 1808
    Other | 3 | 5 | 5 | 13
    Hispanic ethnicity, self-reported: number analyzed (Participants) | 604 | 601 | 603 | 1808
    Hispanic ethnicity, self-reported | 5 | 5 | 10 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Family Member Characteristic -Race/Ethnicity Population: Family Member Race/Ethnicity-excluding missing/withdrawn
  Participants
    Asian: number analyzed (Participants) | 604 | 601 | 603 | 1808
    Asian | 5 | 9 | 3 | 17
    Black or African American: number analyzed (Participants) | 604 | 601 | 603 | 1808
    Black or African American | 92 | 79 | 71 | 242
    White: number analyzed (Participants) | 604 | 601 | 603 | 1808
    White | 504 | 501 | 518 | 1523
    Other: number analyzed (Participants) | 604 | 601 | 603 | 1808
    Other | 2 | 8 | 9 | 19
    Hispanic ethnicity: number analyzed (Participants) | 604 | 601 | 603 | 1808
    Hispanic ethnicity | 3 | 4 | 7 | 14
Severe Depression [Count of Participants; unit: Participants] — Baseline Patient Characteristic- Severe Depression is defined as PHQ-9 score of ≥15 Population: Patient Depressive Symptoms, PHQ-9- The PHQ-9 is a nine-item depression scale with a total score from 0 to 27 with higher scores indicating greater depression severity.
  Participants
    number analyzed (Participants) | 604 | 601 | 603 | 1808
    (all) | 10 | 13 | 12 | 35
Severe Anxiety [Count of Participants; unit: Participants] — Baseline patient characteristic-Severe Anxiety is defined as GAD-7 score of ≥15 Population: Patient Severe Anxiety is defined as GAD-7 score of ≥15 The GAD-7 is a seven-item anxiety scale with a total score from 0 to 21 with higher scores indicating greater anxiety severity.
  Participants
    number analyzed (Participants) | 604 | 601 | 603 | 1808
    (all) | 5 | 12 | 6 | 23
Severe Depression [Count of Participants; unit: Participants] — Baseline Family Characteristic -Severe Depression is defined as PHQ-9 score of ≥15 The PHQ-9 is a nine-item depression scale with a total score from 0 to 27 with higher scores indicating greater depression severity. Population: Family member -Severe Depression is defined as PHQ-9 score of ≥15- excluding missing/withdrawn
  Participants
    number analyzed (Participants) | 604 | 601 | 603 | 1808
    (all) | 8 | 9 | 7 | 24
Severe Anxiety [Count of Participants; unit: Participants] — Baseline Family Characteristic - Severe Anxiety is defined as GAD-7 score of ≥15 The GAD-7 is a seven-item anxiety scale with a total score from 0 to 21 with higher scores indicating greater anxiety severity. Population: Family Member - Severe Anxiety is defined as GAD-7 score of ≥15- excluding missing/withdrawn
  Participants
    number analyzed (Participants) | 604 | 601 | 603 | 1808
    (all) | 6 | 5 | 3 | 14
Oberst Scale, time [Mean (Standard Deviation); unit: units on a scale] — The Oberst Time and Difficulty subscales are two parts of the Oberst Caregiving Burden Scale (OCBS), which measures the perceived time spent and difficulty associated with performing caregiving tasks. Each item is scored on a 5-point response scale. In response to time for each item, the caregiver chooses an amount ranging from no time (score, 1) to a great deal of time (score, 5) spent on tasks related to caregiving. Scores were calculated by averaging across the 15 items of the time and difficulty subscales, thus achieving an average score between 1 and 5 for each subscale. Population: Family member- Oberst Scale, time- excluding missing/withdrawn
  units on a scale
    number analyzed (Participants) | 604 | 601 | 603 | 1808
    (all) | 21.0 (7.3) | 21.0 (7.2) | 20.7 (7.0) | 20.9 (7.1)
Oberst Caregiving Burden Scale, difficulty subscale [Mean (Standard Deviation); unit: units on a scale] — The Oberst Time and Difficulty subscales are two parts of the Oberst Caregiving Burden Scale (OCBS), which measures the perceived time spent and difficulty associated with performing caregiving tasks. Each item is scored on a 5-point response scale. In response to difficulty for each item, the caregiver chooses an amount ranging from not difficult (score, 1) to extremely difficult (score, 5). Scores were calculated by averaging across the 15 items of the time and difficulty subscales, thus achieving an average score between 1 and 5 for each subscale. Population: Family member- Oberst Scale, difficulty- excluding missing/withdrawn
  units on a scale
    number analyzed (Participants) | 604 | 601 | 603 | 1808
    (all) | 15.6 (2.8) | 15.5 (1.8) | 15.6 (1.8) | 15.5 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Short Form Health Survey (SF-36)
Description: The SF-36 is a general population instrument that measures health-related quality of life, mental, physical, and social functioning. It includes one multi-item scale that assesses 8 overall health concepts. These concepts are aggregated into a Physical Component Summary and a Mental Component Summary. The eight domains are combined to reach two summary scores for Physical and Mental Health which are standardized to a mean of 50, with a score above 50 representing better than average and below 50 poorer than average function.
Time Frame: 24 month
Population: Patient & Family Member Outcome Results of SF-36 at 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Screening Only: Screening Only: The patients in this group will receive screening for AD. Patients and family members will receive a letter about how the patient performed on the screening. If they screen positive (e.g. ≤5 on the MIS-T or ≤2 on the Mini-Cog), the patient and family member will receive an infographic and some information about local clinical resources for them to peruse regarding follow-up care. The patient's PCP is also be notified of the screening results via EHR message.
- Screen Plus: Collaborative Care Program: The patients in this group will receive screening for AD, Patients and family members will receive a letter about how the patient performed on the screening. If they screen positive (e.g. ≤5 on the MIS-T or ≤2 on the Mini-Cog), the patient and family member will receive an infographic. Also, the family member will receive two follow-up phone calls. One from the COADS Study Coordinator and one from a care coordinator at the Aging Brain Care Program (ABC). This phone call will include an opportunity for the family to ask questions and a conversation about the program and diagnostic evaluation and management. Dyads have the option to refuse the follow-up visit. The patient's PCP is also be notified of the screening results via EHR message,
Arm/Group | Control | Screening Only | Screen Plus
Number analyzed (Participants) | 1025 | 1023 | 1004
score on a scale
  Family Member- Physical Health Component: number analyzed (Participants) | 505 | 503 | 496
  Family Member- Physical Health Component | 48.4 (9.8) | 47.8 (10.2) | 48.8 (9.4)
  Patient-Physical Health Component: number analyzed (Participants) | 520 | 520 | 508
  Patient-Physical Health Component | 44.7 (11.1) | 44.8 (11.2) | 44.4 (11.1)
  Family Member- Mental Health Component: number analyzed (Participants) | 505 | 503 | 496
  Family Member- Mental Health Component | 54.5 (7.2) | 55.3 (6.7) | 54.7 (7.5)
  Patient-Mental Health Component: number analyzed (Participants) | 520 | 520 | 508
  Patient-Mental Health Component | 54.9 (7.5) | 55.3 (7.4) | 55.3 (7.6)

2. Secondary Outcome: Depressive Symptoms
Description: The investigators will use the Patient Health Questionnaire-9 (PHQ-9) to determine the impact of AD screening on caregivers and patients mood. The PHQ-9 is a nine-item depression scale with a total score from 0 to 27 with higher scores indicating greater depression severity.
  Multi-level mixed effects models will be used to examine differences in PHQ-9 scores for both patients and family members using dyadic analytic approaches. For this aim, we will compare family members in the two screening groups (Screening Only and Screening Plus) to those in the no screening (Control) group. Repeated PHQ-9 scores from both patients and family members will be included as the outcome variables with participant type (patient or family member), group (Screening Only and Screening Plus versus Control), time, and interaction between groups and time as independent variables.
Time Frame: PHQ-9 results for patient & family member at 24 months
Population: PHQ-9 results for patient & family member at 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Screening Only | Screen Plus
Number analyzed (Participants) | 1026 | 1023 | 1006
score on a scale
  Patient 24 Month: number analyzed (Participants) | 520 | 520 | 509
  Patient 24 Month | 2.8 (3.6) | 2.6 (3.8) | 2.9 (3.9)
  Family member 24 Month: number analyzed (Participants) | 506 | 503 | 497
  Family member 24 Month | 2.4 (3.4) | 2.3 (2.9) | 2.2 (3.2)

3. Secondary Outcome: Anxiety Symptoms
Description: The investigators will use the Generalized Anxiety Disorder Scale (GAD-7) to determine the impact of AD screening on caregivers and patients anxiety. The GAD-7 is a seven-item anxiety scale with a total score from 0 to 21 with higher scores indicating greater anxiety severity.
  Multi-level mixed effects models will be used to examine differences in GAD-7 scores for both patients and family members using dyadic analytic approaches. For this aim, we will compare family members in the two screening groups (Screening Only and Screening Plus) to those in the no screening (Control) group. Repeated GAD-7 scores from both patients and family members will be included as the outcome variables with participant type (patient or family member), group (Screening Only and Screening Plus versus Control), time, and interaction between groups and time as independent variables.
Time Frame: 24 month GAD-7 scores for Family members & Patients
Population: 24 month GAD-7 scores for Family members & Patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Screening Only | Screen Plus
Number analyzed (Participants) | 1026 | 1023 | 1006
score on a scale
  Family member: number analyzed (Participants) | 506 | 503 | 497
  Family member | 1.8 (3.0) | 1.6 (2.5) | 1.7 (3.0)
  Patient: number analyzed (Participants) | 520 | 520 | 509
  Patient | 1.7 (2.6) | 1.8 (3.3) | 1.8 (3.0)

4. Secondary Outcome: Caregiving Preparedness
Description: The Preparedness for Caregiving Scale consists of eight items that asks family members how well prepared they believe they are for multiple domains of caregiving. Responses are rated on a 5-point scale with scores ranging from 0 (not at all prepared) to 4 (very well prepared). The scale is scored by calculating the mean of all items answered with a score range of 0 to 4. The higher the score the more prepared the caregiver feels for caregiving; the lower the score, the less prepared the caregiver feels.
  Multi-level mixed effects models will be used to examine differences in Preparedness for Caregiving Scale scores for family members using dyadic analytic approaches. For this aim, we will compare family members in the two screening groups (Screening Only and Screening Plus) to those in the no screening (Control) group. Repeated Preparedness for Care
Time Frame: 24 month
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Screen Plus: Collaborative Care Program: The patients in this group will receive screening for AD, Patients and family members will receive a letter about how the patient performed on the screening. If they screen positive (e.g. ≤5 on the MIS-T or ≤2 on the Mini-Cog), the patient and family member will receive an infographic. Also, the family member will receive two follow-up phone calls. One from the COADS Study Coordinator and one from a care coordinator at the Aging Brain Care Program (ABC). This phone call will include an opportunity for the family to ask questions and a conversation about the program and diagnostic evaluation and management. Dyads have the option to refuse the follow-up visit. The patient's PCP is also be notified of the screening results via EHR message.
Arm/Group | Control | Screening Only | Screen Plus
Number analyzed (Participants) | 505 | 504 | 498
score on a scale | 3.0 (0.7) | 2.9 (0.6) | 2.9 (0.7)

5. Secondary Outcome: Caregiving Self Efficacy
Description: The investigators will use the Revised Scale for Caregiving Self Efficacy to measure the impact of AD screening on caregiver self-efficacy. Respondents rate their degree of self-efficacy on a scale from 0 (absolutely incapable) to 100 (fully capable).
Time Frame: 24 month result for Family member
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Screening Only | Screen Plus
Number analyzed (Participants) | 501 | 504 | 497
score on a scale | 79.1 (15.5) | 79.3 (14.0) | 79.6 (15.0)

ADVERSE EVENTS:
Time Frame: Patient death and hospitalization were collected from EMR quarterly and during participant contact at each study milestone from baseline through 24 month assessment. Family member death and hospitalization were collected during participant contact at study milestones post-baseline at the 6month through 24 month assessment. Patient and Family member risk of severe depression based on post-baseline PHQ-9 and risk of severe anxiety based on post baseline GAD-7 score.
Description: All Cause mortality is the total unique participants all-cause mortality, i.e.. patient and family member mortality combined.
  Serious adverse event include Inpatient Hospitalization or prolongation of existing hospitalization, including patients for all milestones and family member data post-baseline.
  Study risk of severe depression and anxiety were assessed for all patients and family members post-baseline.
Groups:
- Control Patients: The patients in this group will receive no AD screening
- Control Family Member: Represents the Family member of the Control Group patient. The patients in this group will receive no AD screening
- Screening Only Patient: The patients in this group will receive screening for AD. Patients and family members will receive a letter about how the patient performed on the screening. If they screen positive (e.g. ≤5 on the MIS-T or ≤2 on the Mini-Cog), the patient and family member will receive an infographic and some information about local clinical resources for them to peruse regarding follow-up care. The patient's PCP is also be notified of the screening results via EHR message.
- Screening Only Family Member.: Represents the Family member of the Screening only group. The patients in this group will receive screening for AD. Patients and family members will receive a letter about how the patient performed on the screening. If they screen positive (e.g. ≤5 on the MIS-T or ≤2 on the Mini-Cog), the patient and family member will receive an infographic and some information about local clinical resources for them to peruse regarding follow-up care. The patient's PCP is also be notified of the screening results via EHR message.
- Collaborative Dementia Care Program Patients: The patients in this group will receive screening for AD. Patients and family members will receive a letter about how the patient performed on the screening. If they screen positive (e.g. ≤5 on the MIS-T or ≤2 on the Mini-Cog), the patient and family member will receive an infographic. Also, the family member will receive two follow-up phone calls. One from the COADS Study Coordinator and one from a care coordinator at the Aging Brain Care Program (ABC). This phone call will include an opportunity for the family to ask questions and a conversation about the program and diagnostic evaluation and management. Dyads have the option to refuse the follow-up visit. The patient's PCP is also be notified of the screening results via EHR message,
- Collaborative Dementia Care Program Family Member: Represents the Family member of the Collaborative Dementia Care Program. The patients in this group will receive screening for AD. Patients and family members will receive a letter about how the patient performed on the screening. If they screen positive (e.g. ≤5 on the MIS-T or ≤2 on the Mini-Cog), the patient and family member will receive an infographic. Also, the family member will receive two follow-up phone calls. One from the COADS Study Coordinator and one from a care coordinator at the Aging Brain Care Program (ABC). This phone call will include an opportunity for the family to ask questions and a conversation about the program and diagnostic evaluation and management. Dyads have the option to refuse the follow-up visit. The patient's PCP is also be notified of the screening results via EHR message,
Arm/Group | Control Patients | Control Family Member | Screening Only Patient | Screening Only Family Member. | Collaborative Dementia Care Program Patients | Collaborative Dementia Care Program Family Member
All-Cause Mortality (participants affected / at risk) | 24/608 | 8/608 | 19/607 | 9/607 | 12/607 | 5/607
Serious Adverse Events (participants affected / at risk) | 79/608 | 101/608 | 69/607 | 82/607 | 85/607 | 96/607
Other Adverse Events (participants affected / at risk) | 41/608 | 34/608 | 42/607 | 19/607 | 43/607 | 35/607
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Patients (N=608) | Control Family Member (N=608) | Screening Only Patient (N=607) | Screening Only Family Member. (N=607) | Collaborative Dementia Care Program Patients (N=607) | Collaborative Dementia Care Program Family Member (N=607)
Inpatient Hospitalization or prolongation of existing hospitalization (General disorders) | 79 (131) | 101 (159) | 69 (125) | 82 (121) | 85 (134) | 96 (134) — Inpatient Hospitalization of patients and family members either self-reported or discovered through EMR. None were determined protocol related.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Patients (N=608) | Control Family Member (N=608) | Screening Only Patient (N=607) | Screening Only Family Member. (N=607) | Collaborative Dementia Care Program Patients (N=607) | Collaborative Dementia Care Program Family Member (N=607)
Severe Depression Post- Baseline as measured by PHQ-9 (≥15) (Psychiatric disorders) | 26 (48) | 18 (23) | 24 (36) | 11 (15) | 28 (43) | 19 (24) — Severe Depression post-baseline as determined by clinical cut point of score (≥15). Participants were offered resources by PI and no instances were determined as study related.
Severe Anxiety Post-Baseline as measured by GAD-7 (≥15) (Psychiatric disorders) | 15 (19) | 16 (20) | 18 (28) | 8 (10) | 15 (19) | 16 (19) — Severe Anxiety post-baseline as determined by clinical cut point of score (≥15). Participants were offered resources by PI and no instances were determined as study related.

LIMITATIONS AND CAVEATS:
The study staff completed recruitment despite adjustments from Covid-19. Yet, because of the long follow up period, 24-month assessments, we will requested a no cost extension to complete all outcome data collection and analysis. The official award end date was February 28, 2023 and a 12-month NCE extended the project to February 28, 2024, allowing time for data quality check, data analysis and study closeout.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT03300180/Prot_SAP_000.pdf